CLINICAL TRIAL: NCT00189930
Title: A Single-blind, Randomized, Controlled, Phase II Study to Evaluate Immunogenicity and Safety of Two Doses of the MVA-nef HIV Vaccine in HIV-1 Infected Patients With CD4 > 250/µl
Brief Title: An Evaluation of Immunogenicity and Safety of Two Doses of MVA-nef vs. MVA-BN in HIV-1 Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Monika Fluer, Bavarian Nordic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIV-NEF-004; HHSN266200400072C
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infection
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — MVA-HIV-1 nef vaccine; smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): High dose
  Interventions: Biological: MVA-nef
- 2 (Active Comparator): Low dose
  Interventions: Biological: MVA-nef
- 3 (Placebo Comparator)
  Interventions: Biological: IMVAMUNE

INTERVENTIONS:
Biological: MVA-nef — 3 imm.: 5E8_TCID50 MVA-nef, 1E8_TCID50 MVA-nef in non-dominant upper arm
  Arms: 1; 2
Biological: IMVAMUNE — 3 immunizations: 1E8_TCID50 IMVAMUNE
  Arms: 3

SUMMARY:
The objective of the study is to compare two doses of MVA-nef vs. MVA-BN to induce Nef-specific cellular immune response in HIV-1 infected patients

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* HIV-1 infection, as documented by any licensed PCR kit or ELISA (confirmed by an complementary assay e.g. Western blot HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA) at any time prior to study entry.
* Stable on HAART for at least 6 consecutive months prior to study entry (changes of one drug for the another drug due to reasons other than virologic failure are allowed)
* Plasma HIV-1 RNA levels of < 50 copies/ml for at least 6 months prior to study entry (two single blips of up to 200 HIV-1 RNA copies/ml are acceptable if they resolve spontaneously without a change in HAART)
* Plasma HIV-1 RNA levels of < 50 copies/ml at study entry
* CD4 nadir >100
* CD4+ cell counts > 250/µl (one measurement within 4 months prior to study entry and one measurement within screening phase)
* For women, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the volunteer is female and of childbearing potential, she agrees to use an acceptable method of contraception, and not become pregnant for at least 56 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or DepoProvera®) with use of method for a minimum of 30 days prior to vaccination).
* ALT/SGPT, AST/SGOT, and alkaline phosphatase < 3 times institutional upper limit of normal (ULN).
* Urine protein by dipstick or urinalysis < 100mg/dl or <2+ proteinuria
* CBC: Haemoglobin >8 g/dl; White blood cells greater than 2,500 and less than 11,000/mm3; Platelets greater than or equal to 100,000/mm3
* Read, signed and dated informed consent document after being advised of the risks and benefits of the study in a language able to understand, and prior to performance of any study specific procedure
* Cardiac enzymes: within normal range.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Administration of any HIV nef vaccine or vaccinia immunization within the past 5 years.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease on thyroid replacement are not excluded.
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure.
* History or clinical manifestation of clinically significant mental illness or haematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study in the opinion of the investigator.
* ECG with clinical significance (complete left or right bundle branch block, or sustained ventricular arrythmia, or 2 PVCs in a row, or ST elevation consistent with ischemia).
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
* 3 or more of the following risk factors:

  1. High blood pressure requiring therapy.
  2. High blood cholesterol (> 300 mg/dl or ratio LDL/HDL ≥ 3) not induced by the HIV therapy.
  3. Diabetes mellitus or high blood sugar.
  4. He/she has a first degree relative (for example mother, father, brother, or sister) who had a heart condition before the age of 50.
  5. Smoking cigarettes now.
* History of chronic alcohol abuse (40g / day for at least 6 month) and/or intravenous drug abuse (within the past 6 month).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction.
* Acute disease (a moderate or severe illness with or without a fever) at the time of enrolment.
* Any vaccinations with active vaccines within a period starting 30 days prior to administration of the vaccine and ending 30 days after administration of the study vaccine. Any vaccinations with inactive vaccines within a period starting 14 days prior to administration of the vaccine and ending 14 days after administration of the study vaccine.
* Chronic administration (defined as more than 14 days) of immuno- suppressant or immune-modifying drugs during the study period (Corticosteroid nasal sprays are permissible. Subjects who have used topical and inhaled steroids can be enrolled after their therapy is completed).
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at study conclusion.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days or 7 half-lives (whichever is longer) preceding the first dose of the study vaccine, or planned administration of such a drug during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2005-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
T-cell response against MVA-BN and the Nef antigen assessed by intracellular cytokine staining assay (ICS) | 52 Weeks

SECONDARY OUTCOMES:
Occurrence, intensity and relationship of adverse events occurring at any time during the study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Harrer, MD, Principal Investigator — University of Erlangen, Germany
Locations (4):
- Germany (4):
  - University of Erlangen, Erlangen, Bavaria
  - Doctor's Practice, Fürth, Bavaria
  - Doctor's Practice, Munich, Bavaria
  - Doctor's Practice, Nuremberg, Bavaria